CLINICAL TRIAL: NCT06447077
Title: Impact of a Predetermined Day 5 Embryo Transfer Versus a Predetermined Day 6 Embryo Transfer on the Clinical Pregnancy Rate After Intracytoplasmic Sperm Injection (ICSI) Treatment
Brief Title: Impact of a Predetermined Day 5 ET vs. a Predetermined Day 6 ET on Clinical Pregnancy Rate After ICSI Treatment
Status: Recruiting | Type: Observational
Sponsor: Infertility Treatment Center Dortmund (Other)
Collaborators: Fertility Center Dortmund (Unknown); novum - Center for Reproductive Medicine Essen - Duisburg (Unknown); Deutsche Klinik Bad Münder (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Stefan Dieterle, Principal Investigator, University of Witten/Herdecke
Other Study IDs: ET d5 vs d6
Record Dates: First submitted 2024-06-03; First posted 2024-06-06 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Infertility; Reproductive Issues
Keywords: ICSI; Predetermined Day 6 Embryo Transfer; Predetermined Day 5 Embryo Transfer
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 9 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Predetermined embryo transfer on day 5: The control group will include patients who have their oocyte pick-up on a monday (embryo transfer on saturday, day 5), wednesday (embryo transfer on monday, day 5), thursday (embryo transfer on tuesday, day 5), friday (embryo transfer on wednesday, day 5) and saturday (embryo transfer on thursday, day 5).
- Predetermined embryo transfer on day 6: The study group will include patients who have their oocyte pick-up on a tuesday (embryo transfer on monday, day 6).

SUMMARY:
The aim of this prospective multicenter study is to investigate the influence of a predetermined embryo transfer on day 6 compared to a predetermined embryo transfer on day 5. The study population consists of the control group (predetermined embryo transfer on day 5) and the study group (predetermined embryo transfer on day 6). The primary endpoint is the clinical pregnancy rate (detection of a gestational sac) per embryo transfer and the secondary endpoint is the abortion rate per clinical pregnancy. The data from the multicenter study are obtained at three test centers (Fertility Center Dortmund, Fertility Center Essen and Fertility Center Bad Münder).

DETAILED DESCRIPTION:
Since a predetermined embryo transfer on day 5 cannot be performed in some centers on every day of the week (e.g. sunday), some IVF centers perform a predetermined embryo transfer on day 4 or day 6, respepectively. Data for a predetermined embryo transfer on day 4 versus a predetermined embryo transfer on day 5 showed no significant differences regarding clinical pregnancy rates. However, since a day 6 transfer might offer advantages in assessing the development stage, the prolonged culture and transfer on day 6 transfer might be a very promising option.

As of yet, there are no prospective studies in the current literature examining the equivalence of a predetermined embryo transfer on day 6 versus a predetermined embryo transfer on day 5.

The aim of this prospective multicenter study is to investigate the influence of a predetermined embryo transfer on day 6 compared to a predetermined embryo transfer on day 5. The study population consists of the control group (predetermined embryo transfer on day 5) and the study group (predetermined embryo transfer on day 6). The primary endpoint is the clinical pregnancy rate (detection of a gestational sac) per embryo transfer and the secondary endpoint is the abortion rate per clinical pregnancy. The data from the multicenter study are obtained at three test centers (Fertility Center Dortmund, Fertility Center Essen and Fertility Center Bad Münder).

ELIGIBILITY:
Inclusion criteria:

The patients to be included should be ≥18 years old. There is no upper age limit. Only ICSI treatments with a single embryo transfer (SET) should be included. Only the first cycle per patient should be evaluated.

Exclusion criteria:

none

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Female patients seeking ICSI treatment because of male subfertilit
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2024-06-26 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-03 (Estimated)

PRIMARY OUTCOMES:
Clinical pregnancy rate per embryo transfer | 4 weeks after embryo transfer
  Clinical pregnancy rate per embryo transfer (detection of a gestational sac)

SECONDARY OUTCOMES:
Abortion rate per clinical pregnancy | During entire ongoing pregnancy
  Abortion rate per clinical pregnancy (termination of an ongoing clinical pregnancy)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Dieterle, MD, Principal Investigator — University of Witten/Herdecke
Locations (1):
- Infertility treatment center Dortmund, Dortmund, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: No